CLINICAL TRIAL: NCT06289179
Title: Thyroid and Cortisol Hormone Response in Patients With Sepsis Who Attended To Assiut University Hospitals (ICU)
Brief Title: Thyroid and Cortisol Hormone Response to Sepsis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Mahmoud khalf allah Mohamed, Assistant lecturer, Assiut University
Other Study IDs: Thyroid and cortisol in sepsis
Record Dates: First submitted 2024-02-16; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thyroid and cortisol hormone response to sepsis

DETAILED DESCRIPTION:
Sepsis is dysregulated host response to infection that results in life-threatening organ dysfunction. Virtually every body system can be affected by this syndrome to greater or lesser extents.

Endocrine alterations are well characterised in sepsis with variations in circulating blood levels and/or receptor resistance.

In response to any psychological or physical stressor, there is widespread neurohormonal activation to adapt body with the stressor. Production and secretion of stress hormones increase to modulate behaviour Many studies have been performed investigating specific hormonal perturbations such as critical illness-induced corticosteroid insufficiency ,all of which are associated with worse outcomes and poor of body inflammation. However, the endocrine system as a whole has been largely overlooked as a fundamental contributor to the integrated host response to sepsis thyroid axis is affected during sepsis with decreased pituitary release of thyroid stimulating hormone (TSH) and inhibition of the peripheral conversion of thyroxine (T4) by 5-deiodinase to the much more metabolically active triiodothyronine (T3). High cortisol levels also inhibit this enzymatic conversion.

ELIGIBILITY:
Inclusion Criteria:

* The study will include Adults (≥18 years), both genders
* septic patients admitted to critical care unit

Exclusion Criteria:

* thyroid disease
* hypopituitarism
* Addison disease
* Cushing syndrome)

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: include Adults (≥18 years), both genders, admitted to critical care unit with sepsis
  Exclusion patient with Previous diagnosis of endocrinal changes (thyroid dysfunction , hypopituitarism, Addison disease, Cushing syndrome)
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
Pattern of cortisol level and thyroid function response to sepsis in ICU | From time of admission to ICU up to 3rd day after discharge
  Affect of sepsis on hormones at ICU:compare the change of endocrinal hormones ( TSH (mIU/L) .T3(ng/dL) .T4 ( mcg/dL) adrenocorticotropic hormone "ACTH" (pg/mL) , cortisol (µg/dL)) at time of admission, course ICU ,3rd day after discharge

REFERENCES:
- [Background] Silva MH, Araujo MC, Diniz EM, Ceccon ME, Carvalho WB. Thyroid abnormalities in term infants with fungal sepsis. Rev Assoc Med Bras (1992). 2016 Sep;62(6):561-567. doi: 10.1590/1806-9282.62.06.561. PMID 27849234